CLINICAL TRIAL: NCT06002191
Title: Development and Testing of imHere4U: A Digital Suicide Prevention Intervention for Cyberbullied Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Candice Biernesser, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY22070044; K23MH131759 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Psychological Distress; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: The study design is a randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flourish + Questionnaires (Experimental): Participants will be onboarded to Flourish by a research study clinician, following which they will receive a text messaging program for 4 weeks as well as an accompanying resources website. As part of the text messaging program, participants will receive brief questionnaires evaluating their online experiences once every 3 days.
  Interventions: Behavioral: Flourish; Behavioral: Questionnaires of Online Experiences
- Questionnaires Alone (Active Comparator): Participants will be onboarded to a text message program that solely will send participants brief questionnaires evaluating their online experiences once every 3 days.
  Interventions: Behavioral: Questionnaires of Online Experiences

INTERVENTIONS:
Behavioral: Flourish — Flourish is a text messaging program that aims to improve coping following cyberbullying and reduce suicide risk among youth.
  Arms: Flourish + Questionnaires
Behavioral: Questionnaires of Online Experiences — Adolescents will receive brief questionnaires related to their online experiences and the impact those experiences have had on their stress level.

SUMMARY:
The objective of this study is to test the feasibility and preliminary efficacy of Flourish (formerly referred to as imHere4U), a digital suicide prevention intervention for cyberbullied adolescents.

The specific aims are to:

Aim #1: Conduct a randomized controlled trial (RCT) comparing Flourish+Questionnaires vs. Questionnaires Alone among cyberbullied youth at-risk for suicide ages 12-17 (N=80, >35% underserved youth).

H2a. Primary outcome: Feasibility will be evidenced by recruitment/retention rates > 80% and imHere4U engagement > 70%.

H2b. Secondary outcomes: Youth assigned to Flourish+Questionnaires will report improved problem-solving capacity, distress tolerance, and motivation and reduced distress and suicidal ideation than youth assigned to Questionnaires Alone over the 6-month follow-up period.

Exploratory Aim: Examine the feasibility of delivering feedback on online interactions from machine learning algorithms. All youth assigned to Flourish may optionally provide their social media data to receive feedback from machine learning algorithms. H3a. Feedback from algorithms will have high acceptability (identified via qualitative themes and >70% acceptance rates) and usability, defined by mean scores on Post-Study System and Usability Questionnaire (PSSUQ) > 6.

DETAILED DESCRIPTION:
Assessment Visits:

As part of this study, adolescents will participate in four assessment visits at baseline and 4, 12, and 24 weeks following onboarding to the study intervention. Assessments cover a range of topics including mood, anxiety, suicidal thoughts and behaviors, and social media use and experience. At the time of the baseline visit, youth will be selected to receive either Flourish+Questionnaires (intervention condition) or Questionnaires Alone (control condition). Selection will occur through randomization, referring essentially to asking a computer to "flip a coin" to decide which group the participant will be assigned to.

Control Condition: Questionnaires Alone Youth in the control condition will be onboarded to a chatbot by a study clinician. A chatbot refers to an automated intervention that leverages chat-based conversations to communicate intervention content. This chatbot is designed solely to send structured brief questionnaires about online interactions via text messaging. Questionnaires assess the presence of negative/bullying interactions and positive/supportive interactions, once every 3 days. Mirroring the intervention condition, youth will receive this simplified chatbot for 4 weeks. If youth endorse negative/bullying interactions, they will be provided with information for crisis contacts (e.g., crisis hotline information).

Intervention Condition: Flourish Flourish is a chatbot that will aim to improve adolescents' capacity to cope following cyberbullying and reduce their suicidal risk. The duration of Flourish is 4 weeks. Flourish is designed to be self-paced with branching logic, aiming to provide the right type of support at the right time youth need it. Therefore, the frequency with which youth interact with Flourish will differ from person to person. However, participants are expected to interact with Flourish approximately 2-3 times per week.

Onboarding to Flourish. Prior to initiating Flourish, adolescents and their caregivers will participate in a session of approximately 30 minutes with a study clinician in which they will onboard to Flourish. During onboarding, the clinician will orient the adolescent to Flourish and load information onto Flourish that will be available to the adolescent throughout their use of the intervention. This will include personal crisis contacts, such as trusted adults and crisis hotlines they could contact in the event of a crisis, as well as contacts for people they could reach out to for support or distraction outside of a crisis situation, such as a close friend or a family member. Adolescents will additionally enter information to personalize their experience with Flourish, such as entering preferences for coping skills that work best for them. During the onboarding process, caregivers will be provided with resources to respond to cyberbullying as well as information on their child's personal crisis resources.

Questionnaires through Flourish. Youth in the intervention group will receive questionnaires evaluating online experiences mirroring those received by the control group. If adolescents indicate negative interactions, Flourish will automatically launch providing supportive resources including crisis resources. If adolescents indicate supportive interactions (or no interactions), they will be given the option to launch Flourish to practice their coping skills, so they are prepared to respond to future cyberbullying events.

Resource Website for Flourish. Participants receiving Flourish will also have access to an accompanying website. The website will not collect or store any private information from the participant, and the participant will not interact with the website. It is a publicly available website that provides a list of resources participants may use, if needed. For example, this will include youth mental health organizations and organizations that provide education, support, and advocacy for youth who have experienced cyberbullying.

Social Media Data Collection and Feedback. Youth in both groups (Flourish+questionnaires and Questionnaires Alone) will have the option to provide their social media archives as part of the study. Software will strip identifiable information (e.g., names, dates of birth, locations, etc.) to the extent possible from the archives. Archives will be analyzed using software that detects presence of positive and negative social interactions. Those assigned to Flourish+Questionnaires will receive feedback from their online interactions, which is anticipated to help youth gain recognition and awareness of their online environment.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* access to a phone or device capable of text messaging
* past 3-month history of cyberbullying assessed by the cybervictimization subscale of the Traditional Bullying and Cyberbullying Victimization and Perpetration Scale and/or presence of online discrimination measured by a modified version of a discrimination measured developed as part of the Adolescent Brain and Cognitive Development (ABCD) study
* past 3-month history of suicidal risk, including: psychological distress (>13 on the 6-item Kessler Psychological Distress Scale) and/or suicidal ideation or behavior (via the Columbia Suicide Severity Rating Scale)

Exclusion Criteria:

* intellectual challenges, low literacy levels, or other conditions that might inhibit adolescents' ability to effectively engage with Flourish (reported by parents and, if needed, confirmed through the age-appropriate Wechsler Intelligence scale)
* acuity levels suggesting need for a higher level of care (e.g., inpatient hospitalization) or referral for emergency services

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates of eligible participants | Assessed upon recruitment to the study
  Feasibility will be measured through recruitment rates of eligible participants, using a cut-off score of 80% for desirable recruitment rates.
Retention rates of eligible participants | Assessed upon completion of the Week 12 study visits
  Feasibility will be measured through retention rates of eligible participants, using a cut-off score of 80% for desirable retention rates across the 12-week study period.
Level of intervention usage | Assessed upon completion of the 4-week intervention period
  Usage of the intervention will be assessed by engagement with the text messaging intervention one or more times during the study period. A cut-off score of 70% of youth using the intervention one or more times will be used as a minimum requirement for acceptable usage.

SECONDARY OUTCOMES:
Change in psychological distress from baseline to 4 weeks | Assessed at the baseline and Week 4 follow-up assessment visits
  Psychological distress will be measured by the Kessler 6-item psychological distress scale (K6). Total scale scores range from 0 to 24 with higher values indicating higher levels of distress and lower values indicating lower distress.
Change in psychological distress from baseline to 12 weeks | Assessed at the Week 12 follow-up assessment visits
  Psychological distress will be measured by the Kessler 6-item psychological distress scale. Total scale scores range from 0 to 24, higher values indicating higher levels of distress and lower values indicating lower distress.
Change in severity of suicidal ideation and behavior from baseline to 4 weeks | Assessed at baseline and Week 4 follow-up assessment visits
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Change in severity of suicidal ideation and behavior from baseline to 12 weeks | Assessed at baseline and Week 12 follow-up assessment visits
  Severity of suicidal ideation and behavior will be measured with the C-SSRS, an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Change in suicidal ideation from baseline to 4 weeks | Assessed at the baseline and Week 4 assessment visits
  Self-reported suicidal ideation will be measured with the Suicidal Ideation Questionnaire (SIQ). The SIQ has a total score of 0 to 90. Higher scores are indicative of frequent suicidal ideation, and lower scores indicative of infrequent ideation.
Change in suicidal ideation from baseline to 12 weeks | Assessed at the baseline and Week 12 Follow-up assessment visits
  Self-reported suicidal ideation will be measured with the Suicidal Ideation Questionnaire. The SIQ has a total score of 0 to 90. Higher scores are indicative of frequent suicidal ideation, and lower scores indicative of infrequent ideation.

OTHER OUTCOMES:
Change in distress tolerance from baseline to 4 weeks | Assessed at the baseline and Week 4 assessment visits
  Distress tolerance will be measured by the Distress Tolerance Scale. The total score for this scale ranges from 15 to 75 with higher scores indicating higher levels of distress tolerance and lower scores indicating lower distress tolerance.
Change in distress tolerance from baseline to 12 weeks | Assessed at the baseline and Week 12 assessment visit
  Distress tolerance will be measured by the Distress Tolerance Scale. The total score for this scale ranges from 15 to 75 with higher scores indicating higher levels of distress tolerance and lower scores indicating lower distress tolerance.
Change in motivation for help-seeking from baseline to 4 weeks | Assessed at the baseline and Week 4 assessment visits
  Motivation for help-seeking will be measured by Readiness, Importance, and Confidence rulers. This includes three rulers assessing readiness, importance, and confidence in help-seeking following cyberbullying. Scores for each ruler range from 0 (not at all ready) to 10 (very ready).
Change in motivation for help-seeking from baseline to 12 weeks | Assessed at the baseline and Week 12 follow-up assessment visits
  Motivation for help-seeking will be measured by Readiness, Importance, and Confidence rulers. This includes three rulers assessing readiness, importance, and confidence in help-seeking following cyberbullying. Scores for each ruler range from 0 (not at all ready) to 10 (very ready).
Change in social problem-solving from baseline to 4 weeks | Assessed at baseline and Week 4 assessment visits
  Social problem-solving will be measured by the revised, short version of the Social Problem-Solving Inventory. This scale has a total score from 0 to 100 with higher scores indicating more effective problem-solving and lower scores representing a less effective problem-solving.
Change in social problem-solving from baseline to 12 weeks | Assessed at the baseline and Week 12 assessment visits
  Social problem-solving will be measured by the revised, short version of the Social Problem-Solving Inventory. This scale has a total score from 0 to 100 with higher scores indicating more effective problem-solving and lower scores representing a less effective problem-solving.

CONTACTS AND LOCATIONS:
Overall Officials: Candice L Biernesser, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from enrolled participants may be shared with investigators within and outside of the University of Pittsburgh and University of Pittsburgh Medical Center for the purpose of studying cyberbullying or suicide risk among adolescents. Data sharing will be consistent with International Committee of Medical Journal Editors (ICMJE) requirements.
Supporting Information: Study Protocol
Time Frame: These data will be released following acceptance of the project's main outcomes manuscript.
Access Criteria: Data requests may be sent to the PI for review, who will provide data to interested and qualified investigators.